CLINICAL TRIAL: NCT02812459
Title: Short-term Effectiveness of Additional Electrical Stimulation to Exercise Versus Kinesio Taping in Patients With Chronic Low Back Pain: A Randomized Controlled Trial
Brief Title: Effectiveness of Electrical Stimulation or Kinesio Taping on Recovery Disability in Low Back Pain
Acronym: ELECBACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Encarnación Aguilar Ferrandiz, Lecturer, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ELECBACK_KT
Record Dates: First submitted 2016-06-16; First posted 2016-06-24 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Chronic Low Back Pain
Keywords: Electrical Stimulation Therapy; Kinesio taping; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kinesio taping plus exercise (Experimental): Kinesio taping application for low back plus back exercises.This protocol will be administered three a week for 4 weeks.
  Interventions: Other: Kinesio taping
- Electrical stimulation plus exercise (Active Comparator): Electrical stimulation for control pain applied in low back plus exercises.This protocol will be administered three a week for 4 weeks.
  Interventions: Other: Electrical Stimulation

INTERVENTIONS:
Other: Kinesio taping — Kinesio taping is a new taping modality which act diminishing pain.
  Arms: Kinesio taping plus exercise
Other: Electrical Stimulation — Electrical stimulation therapy is a electrical current that allow patients diminish pain.
  Arms: Electrical stimulation plus exercise

SUMMARY:
The purpose of this study is to analyze the effectiveness of electrical stimulation and kinesio taping in combination with exercise in People with Chronic Low Back Pain

ELIGIBILITY:
Inclusion Criteria:

1. LBP for three months or more;
2. age between 25 and 65 years;
3. a score of four points or more on the Roland Morris Disability Questionnaire;
4. not currently receiving physical therapy.

Exclusion Criteria:

1. the presence of lumbar stenosis;
2. any clinical signs of radiculopathy;
3. a diagnosis of spondylolisthesis;
4. a diagnosis of fibromyalgia;
5. treatment with corticosteroid or oral medication within the past two weeks;
6. a history of spinal surgery;
7. disease of the central or peripheral nervous system.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-06; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Roland Morris Disability Questionnaire (RMDQ) at one month. | 4 weeks
  The Roland Morris disability questionnaire is a self-administered disability measurement scored on a 24-point scale from 0 = no disability to 24 = severe disability

SECONDARY OUTCOMES:
Change from baseline Oswestry Disability Index (ODI) at one month. | 4 weeks
  The Oswestry disability index evaluates daily life activity limitations in 10 dimensions, each scored on a 6-point scale (0-5 points); the total points scored are expressed as a percentage, used to classify individuals as minimally disabled (0-10%), moderately disabled (20-40%), severely disabled (40-60%), crippled (60-80%), or bedbound (80-100%).
Change from baseline Visual Analogue Scale (VAS) at one month | 4 weeks
  The visual analogue scale for pain intensity ranged from 0 = no pain to 10 = worst imaginable pain
Change from baseline Tampa Scale for Kinesiophobia (TSK) at one month | 4 weeks
  The Tampa Scale for Kinesiophobia comprises 17 items on the fear of movement or recurrent lesion, each scored on a 4-point Likert scale from "completely disagree" to "completely agree".
Change from baseline Pressure pain thresholds (PPT) at one month | 4 weeks
  Examination of PPT will be performed with the use of an Algometer. According to International Association for the Study of Pain, PPT is the smallest stimulus causing the feeling of pain (International Association for the Study of Pain, Subcommittee on Taxonomy, 1986). The examination will carried out twice in the same places, on the left and right sides following the protocol described by Sipko et al.2013: musculus erector spinae - at the level of L2, 3 cm away from the interspinous line; musculus gluteus medius - between the greater trochanter and iliac crest sideways; musculus triceps surae - the transition of the belly of the muscle into the tendon; and musculus tibialis anterior - one-third of the upper shank, at the front.
Change from baseline Mechanosensitive/the Seated Slump Test neurodynamic testing at one month | 4 weeks
  The subject will be positioned in an erect sitting position on an examination plinth with the popliteal creases just off the edge of the plinth. The subject will be asked to sit in a slouched position. After, the subject will be asked to actively flex the cervical spine as far as comfortably possible. After, the subject's ankle will be then passively dorsiflexed to slight resistance, while the knee is slowly passively extended.The knee will be extended until the subject reports onset of neural-mediated symptoms.The degree of knee extension will be measured with a large universal goniometer.
Change from baseline Mechanosensitive/straight-leg raise neurodynamic testing at one month | 4 weeks
  The subject will be positioned in supine with standardized head support. After the test will be performed with the ankle in neutral position and with 30º of ankle flexion. The hip will be flexed with the knee extended until the subject reports onset of neural-mediated symptoms. The degree of hip flexion will be measured with a large universal goniometer.
Change from baseline Anxiety and depression measures at one month | 4 weeks
  Beck questionnaire
Change from baseline Quality of Sleep at one month | 4 weeks
  Pittsburgh questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: María Encarnación Aguilar-Ferrándiz, Principal Investigator — Deparment of Physical Therapy. University of Granada
Locations (1):
- Adelaida Mª Castro Sánchez, Almería, Spain

REFERENCES:
- [Background] Boyd BS, Wanek L, Gray AT, Topp KS. Mechanosensitivity of the lower extremity nervous system during straight-leg raise neurodynamic testing in healthy individuals. J Orthop Sports Phys Ther. 2009 Nov;39(11):780-90. doi: 10.2519/jospt.2009.3002. PMID 19881004
- [Background] Fritz JM, Irrgang JJ. A comparison of a modified Oswestry Low Back Pain Disability Questionnaire and the Quebec Back Pain Disability Scale. Phys Ther. 2001 Feb;81(2):776-88. doi: 10.1093/ptj/81.2.776. PMID 11175676
- [Background] Sipko T, Kuczynski M. Intensity of chronic pain modifies postural control in low back patients. Eur J Pain. 2013 Apr;17(4):612-20. doi: 10.1002/j.1532-2149.2012.00226.x. PMID 23065907
- [Result] Deyo RA, Weinstein JN. Low back pain. N Engl J Med. 2001 Feb 1;344(5):363-70. doi: 10.1056/NEJM200102013440508. No abstract available. PMID 11172169
- [Result] Ekman M, Johnell O, Lidgren L. The economic cost of low back pain in Sweden in 2001. Acta Orthop. 2005 Apr;76(2):275-84. doi: 10.1080/00016470510030698. PMID 16097556
- [Result] Melloh M, Elfering A, Stanton TR, Kaser A, Salathe CR, Barz T, Roder C, Theis JC. Who is likely to develop persistent low back pain? A longitudinal analysis of prognostic occupational factors. Work. 2013 Jan 1;46(3):297-311. doi: 10.3233/WOR-131672. PMID 24004738
- [Result] Hallegraeff JM, Krijnen WP, van der Schans CP, de Greef MH. Expectations about recovery from acute non-specific low back pain predict absence from usual work due to chronic low back pain: a systematic review. J Physiother. 2012;58(3):165-72. doi: 10.1016/S1836-9553(12)70107-8. PMID 22884183
- [Result] Costa Lda C, Maher CG, McAuley JH, Hancock MJ, Herbert RD, Refshauge KM, Henschke N. Prognosis for patients with chronic low back pain: inception cohort study. BMJ. 2009 Oct 6;339:b3829. doi: 10.1136/bmj.b3829. PMID 19808766
- [Result] Added MA, Costa LO, de Freitas DG, Fukuda TY, Monteiro RL, Salomao EC, de Medeiros FC, Costa Lda C. Kinesio Taping Does Not Provide Additional Benefits in Patients With Chronic Low Back Pain Who Receive Exercise and Manual Therapy: A Randomized Controlled Trial. J Orthop Sports Phys Ther. 2016 Jul;46(7):506-13. doi: 10.2519/jospt.2016.6590. Epub 2016 Jun 6. PMID 27266883
- [Result] Forozeshfard M, Bakhtiary AH, Aminianfar A, Sheikhian S, Akbarzadeh Z. Short term effects of kinesio taping on pain and functional disability in young females with menstrual low back pain: A randomised control trial study. J Back Musculoskelet Rehabil. 2016 Nov 21;29(4):709-715. doi: 10.3233/BMR-160673. PMID 26966819
- [Result] Luz Junior MA, Sousa MV, Neves LA, Cezar AA, Costa LO. Kinesio Taping(R) is not better than placebo in reducing pain and disability in patients with chronic non-specific low back pain: a randomized controlled trial. Braz J Phys Ther. 2015 Nov-Dec;19(6):482-90. doi: 10.1590/bjpt-rbf.2014.0128. Epub 2015 Oct 9. PMID 26647750
- [Result] Kelle B, Guzel R, Sakalli H. The effect of Kinesio taping application for acute non-specific low back pain: a randomized controlled clinical trial. Clin Rehabil. 2016 Oct;30(10):997-1003. doi: 10.1177/0269215515603218. Epub 2015 Aug 27. PMID 26316553
- [Result] Hagen L, Hebert JJ, Dekanich J, Koppenhaver S. The effect of elastic therapeutic taping on back extensor muscle endurance in patients with low back pain: a randomized, controlled, crossover trial. J Orthop Sports Phys Ther. 2015 Mar;45(3):215-9. doi: 10.2519/jospt.2015.5177. Epub 2015 Feb 13. PMID 25679343
- [Result] Kachanathu SJ, Alenazi AM, Seif HE, Hafez AR, Alroumim MA. Comparison between Kinesio Taping and a Traditional Physical Therapy Program in Treatment of Nonspecific Low Back Pain. J Phys Ther Sci. 2014 Aug;26(8):1185-8. doi: 10.1589/jpts.26.1185. Epub 2014 Aug 30. PMID 25202177
- [Result] Alvarez-Alvarez S, Jose FG, Rodriguez-Fernandez AL, Gueita-Rodriguez J, Waller BJ. Effects of Kinesio(R) Tape in low back muscle fatigue: randomized, controlled, doubled-blinded clinical trial on healthy subjects. J Back Musculoskelet Rehabil. 2014;27(2):203-12. doi: 10.3233/BMR-130437. PMID 24284272
- [Result] Elserty N, Kattabei O, Elhafez H. Effect of Fixed Versus Adjusted Transcutaneous Electrical Nerve Stimulation Amplitude on Chronic Mechanical Low Back Pain. J Altern Complement Med. 2016 Jul;22(7):557-62. doi: 10.1089/acm.2015.0063. Epub 2016 May 4. PMID 27144300
- [Result] Jauregui JJ, Cherian JJ, Gwam CU, Chughtai M, Mistry JB, Elmallah RK, Harwin SF, Bhave A, Mont MA. A Meta-Analysis of Transcutaneous Electrical Nerve Stimulation for Chronic Low Back Pain. Surg Technol Int. 2016 Apr;28:296-302. PMID 27042787
- [Result] Hicks GE, Sions JM, Velasco TO, Manal TJ. Trunk Muscle Training Augmented With Neuromuscular Electrical Stimulation Appears to Improve Function in Older Adults With Chronic Low Back Pain: A Randomized Preliminary Trial. Clin J Pain. 2016 Oct;32(10):898-906. doi: 10.1097/AJP.0000000000000348. PMID 26736024
- [Result] Pivec R, Minshall ME, Mistry JB, Chughtai M, Elmallah RK, Mont MA. Decreased Opioid Utilization and Cost at One Year in Chronic Low Back Pain Patients Treated with Transcutaneous Electric Nerve Stimulation (TENS). Surg Technol Int. 2015 Nov;27:268-74. PMID 26680409
- [Result] Gladwell PW, Badlan K, Cramp F, Palmer S. Problems, Solutions, and Strategies Reported by Users of Transcutaneous Electrical Nerve Stimulation for Chronic Musculoskeletal Pain: Qualitative Exploration Using Patient Interviews. Phys Ther. 2016 Jul;96(7):1039-48. doi: 10.2522/ptj.20150272. Epub 2015 Dec 17. PMID 26678446
- [Result] Frahm KS, Hennings K, Vera-Portocarrero L, Wacnik PW, Morch CD. Nerve Fiber Activation During Peripheral Nerve Field Stimulation: Importance of Electrode Orientation and Estimation of Area of Paresthesia. Neuromodulation. 2016 Apr;19(3):311-8. doi: 10.1111/ner.12371. Epub 2015 Nov 19. PMID 26586248
- [Derived] Aguilar-Ferrandiz ME, Mataran-Penarrocha GA, Tapia-Haro RM, Castellote-Caballero Y, Marti-Garcia C, Castro-Sanchez AM. Effects of a supervised exercise program in addition to electrical stimulation or kinesio taping in low back pain: a randomized controlled trial. Sci Rep. 2022 Jul 6;12(1):11430. doi: 10.1038/s41598-022-14154-5. PMID 35794120